CLINICAL TRIAL: NCT03249142
Title: A Multicentre Feasibility Randomized Study of Anti-PD-L1 Durvalumab (MEDI4736) With or Without Anti-CTLA-4 Tremelimumab in Patients With Ovarian, Fallopian Tube or Primary Peritoneal Adenocarcinoma, Treated With a First-line Neo-adjuvant Strategy
Brief Title: Immunotherapy With Neo-adjuvant Chemotherapy for OVarian Cancer
Acronym: INeOV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GINECO-OV127b
Record Dates: First submitted 2017-08-04; First posted 2017-08-15 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Anti-PD-L1; Anti-CLA-4; Neo-adjuvant
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A Durvalumab/chemotherapy association (Experimental)
  Interventions: Drug: ARM A Durvalumab/chemotherapy association
- ARM B Durvalumab/Tremelimumab/chemotherapy association (Experimental)
  Interventions: Drug: ARM B Durvalumab/Tremelimumab/chemotherapy association

INTERVENTIONS:
Drug: ARM A Durvalumab/chemotherapy association — NEO-ADJUVANT Cycle 1 : carboplatin AUC 5 IV + paclitaxel 175 mg/m² IV alone (day1), every 3 weeks Cycle 2 : carboplatin AUC 5 IV + paclitaxel 175 mg/m² IV + durvalumab 1125 mg IV (day1) Cycle 3 : carboplatin AUC 5 IV + paclitaxel 175 mg/m² IV + durvalumab 1125 mg IV (day1)
  ADJUVANT :
  1. If complete surgical resection at interval debulking surgery : 3 cycles of durvalumab 1125 mg IV + carboplatin AUC 5 IV + paclitaxel 175 mg/m² IV at day1, every 3 weeks.
  2. If residual tumor at interval debulking surgery : the tremelimumab 75 mg IV will be added to the durvalumab-chemotherapy combination at day 1 of cycle 2 before a salvage surgery. Durvalumab 1125 mg IV (with one cycle of tremelimumab 75 mg IV post S3) will be pursued in maintenance treatment, up to 1 year or until disease progression, unacceptable toxicity or patient withdrawn.
  Arms: ARM A Durvalumab/chemotherapy association
Drug: ARM B Durvalumab/Tremelimumab/chemotherapy association — NEO-ADJUVANT Cycle 1 : carboplatin AUC 5 IV + paclitaxel 175 mg/m² IV alone (day1), every 3 weeks Cycle 2 : carboplatin AUC 5 IV + paclitaxel 175 mg/m² IV + durvalumab 1125 mg IV + tremelimumab 75 mg IV (day1) Cycle 3 : carboplatin AUC 5 IV + paclitaxel 175 mg/m² IV + durvalumab 1125 mg IV (day1)
  ADJUVANT :
  1. If complete surgical resection at interval debulking surgery : 3 cycles of durvalumab 1125 mg IV + carboplatin AUC 5 IV + paclitaxel 175 mg/m² IV at day1, every 3 weeks.
  2. If residual tumor at interval debulking surgery : patients will be treated according to investigator choice.
  Arms: ARM B Durvalumab/Tremelimumab/chemotherapy association

SUMMARY:
This is a randomized, open, comparative, multi-centre study which will recruit up to 66 patients. The objective is mainly to explore the safety and feasibility in neo-adjuvant first-line ovarian cancer (including patients with primary peritoneal or fallopian tube adenocarcinoma) of various combinations of durvalumab with chemotherapy with or without tremelimumab.

DETAILED DESCRIPTION:
The schedule is the following:

• In a first step a run-in phase of 6 patients will be conducted to test the safety and feasibility of the combination of durvalumab with standard carboplatin-paclitaxel chemotherapy.

Cycle 1 : chemotherapy alone (day1) Cycle 2 : chemotherapy + durvalumab (day1) Cycle 3 : chemotherapy + durvalumab (day1)

• In a second step, if first-step was found feasible, a run-in phase of 6 patients will be conducted to test the safety and feasibility of the combination of durvalumab plus tremelimumab with standard carboplatin-paclitaxel chemotherapy.

Cycle 1 : chemotherapy alone (day1) Cycle 2 : chemotherapy + durvalumab + tremelimumab (day1) Cycle 3 : chemotherapy + durvalumab (day1)

* After the run-in phase, patients will be randomized in a ratio 1:1 between those included in the durvalumab-chemotherapy expansion phase (arm A) and those included in the durvalumab + tremelimumab-chemotherapy expansion phase (arm B).
* This study will also allow to explore the feasibility of a salvage therapy personalized according to the results of interval surgery and type of previous neo-adjuvant therapy.

  1. In those patients who achieved a complete surgical resection at interval debulking surgery, adjuvant treatment will include 3 cycles of durvalumab + chemotherapy and then a follow-up period.
  2. In patients with residual tumor at interval debulking surgery, salvage therapy will depend on the initial treatment arm allocated.

     1. In arm A, the tremelimumab will be added to the durvalumab-chemotherapy combination at day 1 of cycle 2 before a salvage surgery. Durvalumab (with one cycle of tremelimumab post S3) will be pursued in maintenance treatment, up to 1 year or until disease progression, unacceptable toxicity or patient withdrawn.
     2. In arm B, the therapy will be according to the Investigator choice and managed according to local practice.

ELIGIBILITY:
Inclusion Criteria:

I-1 Female patients must be ≥ 18 years of age. I-2 Signed informed consent and ability to comply with treatment and follow-up. I-3 Patients with newly histologically confirmed epithelial ovarian cancer (or fallopian tube or primary peritoneal adenocarcinoma).

I-4 Advanced FIGO stage IIIC to IV. I-5 Patients for whom primary debulking surgery has been denied after an evaluation through laparoscopy or laparotomy.

I-6 Patient for whom a neo-adjuvant strategy has been planned. I-7 Interval between diagnosis and enrolment (informed consent signed) ≤ 8 weeks.

I-8 Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1. I-9 Geriatric vulnerability score (GVS) < 3 for patients ≥ 70 years. I-10 Adequate organ and bone marrow function. I-11 Patients not receiving anticoagulant medication who have an International Normalized Ratio (INR) ≤ 1.5 and an Activated ProThrombin Time (aPTT) ≤ 1.5 x ULN. The use of full-dose oral or parenteral anticoagulants is permitted as long as the INR or aPTT is within therapeutic limits (according to site medical standard) and if the patient is on a stable dose of anticoagulants for at least two weeks at the time of randomization.

I-12 As this study will include patients in France, a subject will be eligible for randomization in this study only if either affiliated to, or a beneficiary of, a social category.

Exclusion Criteria:

E-1 Other malignancy within the last 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS).

E-2 Major surgical procedure (defined by the resection of at least one organ including ovary) within 28 days prior to the first dose.

E-3 Any concurrent chemotherapy, investigational product, biological, or hormonal therapy for cancer treatment.

E-4 Previous treatment with immunotherapy, including, but not limited to, anti-CTLA-4, anti-PD-1, anti-PD-L1, or anti-PD-L2 antibodies, or therapeutic anticancer vaccine.

E-5 Active or prior documented autoimmune or inflammatory disorders The following are exceptions to this criterion:

1. Patients with vitiligo or alopecia,
2. Patients with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement or psoriasis not requiring systemic treatment.

E-6 Current/prior immunosuppressive medication ≤ 14 days before first durvalumab and tremelimumab dose (including, but not limited to, prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF] agents) within 2 weeks prior to Cycle 1, Day 1, or anticipated requirement for systemic immunosuppressive medications during the trial.

E-7 Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV). Patients with active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C. Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible.

E-8 Uncontrolled diabetes mellitus, uncontrolled hypothyroidism. E-9 Treatment with systemic immunostimulatory agents (including but not limited to interferon-alpha (IFN-α) and interleukin-2 (IL-2) within 4 weeks or five half- lives of the drug (whichever is shorter) prior to Cycle 1, Day 1.

E-10 History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis. Radiation pneumonitis in the radiation field (fibrosis) detected on screening chest CT scan is permitted.

E-11 Signs or symptoms of infection within 2 weeks prior to Cycle 1, Day 1. E-12 Administration of a live, attenuated vaccine within 4 weeks prior to Cycle 1, Day 1 or anticipation that such a live attenuated vaccine will be required during the study. Influenza vaccination should be given during influenza season only (example approximately October to March in the Northern Hemisphere). Patients must not receive live, attenuated influenza.

E-13 Current or recent (within 10 days prior to randomization) chronic use of aspirin > 325 mg/day.

E-14 Prior history of hypertensive crisis (CTC-AE grade 4) or hypertensive encephalopathy.

E-15 Inadequately controlled HTN (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg on antihypertensive medications).

E-16 Clinically significant (e.g. active) cardiovascular disease, including:

1. Myocardial infarction or unstable angina within ≤ 6 months of randomization,
2. New York Heart Association (NYHA) ≥ grade 2 congestive heart failure (CHF),
3. Poorly controlled cardiac arrhythmia despite medication (patients with rate controlled atrial fibrillation are eligible),
4. Peripheral vascular disease grade ≥ 3 (e.g. symptomatic and interfering with activities of daily living [ADL] requiring repair or revision).

E-17 Previous Cerebro-Vascular Accident (CVA), Transient Ischemic Attack (TIA) or Sub-Arachnoids Hemorrhage (SAH) within 6 months prior to randomization.

E-18 History or evidence of hemorrhagic disorders within 6 months prior to randomization.

E-19 Evidence of bleeding diathesis or significant coagulopathy (in the absence of coagulation).

E-20 History or clinical suspicion of brain metastases or spinal cord compression unless asymptomatic, treated, and stable off steroids and anti-convulsants for at least 1 month prior to entry.

E-21 History or evidence upon neurological examination of central nervous system (CNS) disease, unless adequately treated with standard medical therapy (e.g. uncontrolled seizures).

E-22 Pre-existing motor or sensory neurotoxicity (grade > 1). E-23 Significant traumatic injury within 4 weeks prior to randomization. E-24 Non-healing wound, active ulcer or bone fracture. Patients with granulating incisions healing by secondary intention with no evidence of facial dehiscence or infection are eligible but require 3 weekly wound examinations.

E-25 Current, clinically relevant bowel obstruction, including sub-occlusive disease, related to underlying disease.

E-26 Previous allogeneic bone marrow transplant or previous solid organ transplantation.

E-27 Patients with evidence of abdominal free air not explained by paracentesis or recent surgical procedure.

E-28 Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment related complications.

E-29 Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential (< 2 years after last menstruation and not surgically sterile) who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period.

E-30 History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.

E-31 Known hypersensitivity or allergy to biopharmaceuticals or to any component of the durvalumab or tremelimumab formulations.

E-32 Known hypersensitivity reaction or allergy to drugs chemically related to carboplatin, paclitaxel, or their excipients that contraindicates the subject's participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Toxicity after neo-adjuvant treatment | At the end of cycle 3 (each cycle is 21 days)
  frequency of adverse events according to CTCAE v4.03 criteria

SECONDARY OUTCOMES:
Toxicity after adjuvant treatment | At the end of cycle 6 (each cycle is 21 days)
Toxicity after maintenance therapy | Up to 18 months
Safety after interval debulking surgery | Up to 6 months
  adverse events according to the Clavien-Dindo classification
Progression Free Survival (PFS) based on investigator assessment using the RECIST version 1.1 | From date of randomisation until the date of progression or death, which ever occurs earlier, assessed up to 36 months
Sugarbaker Peritoneal Index Score (PCI) | Up to 6 months
Time to start of first subsequent therapy or death | Up to 36 months
overall survival | from date of randomisation to death, assessed up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra LEARY, MD, PhD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (11):
- France (11):
  - Institut Ste Catherine, Avignon
  - Institut Bergonié, Bordeaux
  - ICM Val d'Aurelle, Montpellier
  - Groupe confluent, Nantes
  - HEGP, Paris
  - Hôpital Cochin, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut René Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No